CLINICAL TRIAL: NCT06186141
Title: A Comparison of Nausea and Vomiting in Postoperative Paediatric Patients With Patient-controlled Analgesia (PCA): Morphine vs Oxycodone (POPCORN)
Brief Title: Nausea and Vomiting in Postoperative Paediatric Patients With Patient-Controlled Analgesia (PCA): Morphine vs Oxycodone
Acronym: POPCORN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91523
Record Dates: First submitted 2023-12-16; First posted 2023-12-29 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Patient-Controlled Analgesia
Keywords: Post-operative Pain; Paediatric; Patient-controlled analgesia; Paediatric analgesia; Post-operative; Embedded clinical trials
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Oxycodone

STUDY DESIGN:
Intervention Model Description: This is a single site randomised embedded trial comparing the side effects of two standard intravenous opioid PCAs, namely morphine and oxycodone. There are two treatment arms, namely morphine and oxycodone, with patients randomised to each arm. Apart from the consent and randomisation process there will be no change to current pre-existing practices for PCAs and patient care.
Masking Description: The study will not be blinded due to the need for opioid syringes to be readily identifiable on the ward.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous (IV) Morphine Patient controlled analgesia (PCA) (Active Comparator): Morphine PCA IV 20mcg/kg bolus to a maximum of 1mg with a 5-minute lockout- as per current RCH Children's Pain Management Service (CPMS) dosing and use.
  Interventions: Drug: Morphine
- IV Oxycodone PCA (Active Comparator): Oxycodone PCA IV 20mcg/kg bolus to a maximum of 1mg with a 5-minute lockout- as per current RCH Children's Pain Management Service (CPMS) dosing and use.
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Morphine — Intravenous (IV) delivery via Patient Controlled Analgesia device (PCA) 20mcg/kg bolus to a maximum of 1mg with a 5-minute lockout
  Arms: Intravenous (IV) Morphine Patient controlled analgesia (PCA)
Drug: Oxycodone — Intravenous (IV) delivery via Patient Controlled Analgesia device (PCA) 20mcg/kg bolus to a maximum of 1mg with a 5-minute lockout
  Other Names: Oxycodone Juno; Oxycodone HCI Medsurge
  Arms: IV Oxycodone PCA

SUMMARY:
POPCORN trial will compare the side effects and effectiveness of Morphine versus Oxycodone medication when prescribed for use as patient controlled analgesia (PCA) for pain relief for paediatric patients after-surgery. This trial is embedded into routine patient care using the hospital electronic medical record (EMR). Participants will be randomly assigned to either medication after they enrol in the study.

The main questions the POPCORN trial aims to answer are:

* 1. Is there a difference in the usage of medication to treat nausea and vomiting for those who received oxycodone PCA versus morphine PCA for post-surgery pain relief?
* 2. Is there a difference in side effects or pain relief needed between the two groups?

Study activities are as follows:

* Participants enrolled to study during their pre-operative consultation
* Participants are randomly assigned to morphine or oxycodone
* No further study-specific activities expected from participant after enrolment and randomisation
* Participant receives routine medical care as planned
* Clinicians record assessments as per routine care in electronic medical record (EMR)
* EMR data are extracted as trial data

DETAILED DESCRIPTION:
Morphine and oxycodone are commonly used intravenous (IV) opioids in adult and paediatric post-operative patients. Traditionally, morphine has been preferentially prescribed with PCA. However, IV oxycodone is rapidly becoming more popular. Despite systematic reviews describing their use within the adult population, very little is known about the comparative side-effect profiles of morphine versus oxycodone within the paediatric post-operative population. Both options are currently in use and considered standard of care at The Royal Children's Hospital (RCH), Melbourne, Australia. However, there is limited literature to support a clinician's choice between IV oxycodone PCA versus IV morphine PCA.

The aim of this embedded randomized controlled trial is to compare the side-effect profile of IV oxycodone PCA to IV morphine PCA in post-operative paediatric patients.

This is a single site, randomised, embedded trial with two intervention arms, namely IV morphine PCA and IV oxycodone PCA. The study will not be blinded due to the need for opioid syringes to be readily identifiable on the ward. Apart from the consent and randomisation process, there will be no change to current pre-existing practices around PCA use and patient care. Adopting a health informatics approach; patient identification, consent, randomization and reporting of outcomes will be embedded within the EMR.

The primary objective is to compare antiemetic use between the two intervention arms. The secondary objectives will be a comparison of PCA side effects, efficacy and opioid use between the two arms. Outcome data must be what is already recorded as part of usual clinical care within the EMR including: antiemetic administration, respiratory depression (new oxygen and/or high dose naloxone use), urinary retention (need for in-dwelling catheter insertion), constipation (medication laxative administration), itch (RCH Itch Score (0-4 Likert scale)), nausea and vomiting, sedation (0-4 University of Michigan Scoring System), pain (Wong-Baker FACES Pain Rating Scale/Visual Analogue Scale (VAS 0-10) and total opioid consumption (mg/kg/day).

ELIGIBILITY:
Inclusion Criteria:

* Postoperative patients who are appropriate for a PCA including those aged 6 and above and up to age 18 years.
* Those deemed appropriate for either morphine or oxycodone by their treating anaesthetist.
* American Society of Anaesthesiologists (ASA) score 1-3 inclusive
* Those whose parents or legal guardians have provided informed consent on the patient's behalf.

Exclusion Criteria:

* Any patients with an allergy, hypersensitivity, or contraindication to morphine or oxycodone.
* Patients in the age group with significant intellectual disability or physical incapacity rendering them incapable of using the PCA device
* ASA score 4 or above
* Inability or unwillingness of parent or legal guardian to provide informed consent for the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 690 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2027-03-19 (Estimated)

PRIMARY OUTCOMES:
Antiemetic use | From PCA attachment to 72 hours or 4 hours after ceasing PCA, whichever is first.
  Prescription incidence and administration of any of the following to participant: Granisetron, Ondansetron, Droperidol, Metoclopramide, Cyclizine, Dexamethasone, and Promethazine

SECONDARY OUTCOMES:
Incidence of Respiratory Depression | The time at which the PCA is first attached to the child and either up to 72 hours or 4 hours after ceasing PCA, whichever is first.
  Measured as any new oxygen and/or high dose naloxone use (10mcg/kg to max of 400mcg). This will exclude administration of low dose naloxone when used to manage incidence of itch.
Incidence of Urinary Retention | From PCA attachment to 72 hours or 4 hours after ceasing PCA, whichever is first.
  Indicated by need for an in-dwelling catheter (IDC) insertion
Reports of Itch | From PCA attachment to 72 hours or 4 hours after ceasing PCA, whichever is first.
  Measured using RCH Itch Score (0-4 Likert scale) where a higher score indicates worse pruritus/itch.
  0=comfortable, no itch, 1=itches a little, doesn't interfere with activity, 2= itches more, sometimes interferes with activity, 3= itches a lot, difficult to be still/concentrate, 4= itches most terribly, impossible to sit still/concentrate
Reports of Nausea | From PCA attachment to 72 hours or 4 hours after ceasing PCA, whichever is first.
  Measured via 0-10 visual analogue scale (VAS) scale Nausea will be measured using the nausea scale (0-10 Baxter Retching Faces scale / VAS)
Sedation levels | From PCA attachment to 72 hours or 4 hours after ceasing PCA, whichever is first.
  Measured via University of Michigan Scoring System (0-4 scale) where a higher score indicates higher sedation level.
  0= awake and alert, 1= minimally sedated, 2=moderately sedated, 3=deep sedation, 4=unrousable
Incidence of Constipation | From PCA attachment to 72 hours or 4 hours after ceasing PCA, whichever is first.
  Recorded laxative administered is indicative. Medication laxatives only, no food laxatives.
Reported pain levels | From PCA attachment to 72 hours or 4 hours after ceasing PCA, whichever is first.
  Measured via Wong-Baker FACES Pain Rating Scale or Visual Analogue Scale (0-10) higher is more pain. If both a pain scale and a rating are reported but don't align the higher of the two will be used.
Total opioid consumption | From PCA attachment to 72 hours or 4 hours after ceasing PCA, whichever is first.
  All opioids administered, including any background infusions are accurately documented in the EMR. Total opioid administered will be calculated from the EMR. The total morphine equivalent dose will be calculated.
Incidence of Vomiting | From PCA attachment to 72 hours or 4 hours after ceasing PCA, whichever is first.
  Incidence of vomiting will be measured using the documentation of number of vomiting episodes. This will be reported for each day over the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Sue May Koh, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- The Royal Children's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Beginning 12 months following analysis and article publication, the following will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by the Murdoch Children's Research Institute's (MCRI's) independent data use review committee (not including trial sponsor-investigator) and who accept MCRI's conditions, under a collaborator agreement, for accessing participant data after de-identification (text, tables, figures, and appendices) that underlies reported results, along with trial protocol, Statistical Analysis Plan (SAP) and Participant Information and Consent Forms (PICF).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 12 months following analysis and publication of the primary outcome
Access Criteria: Requests for access to previously published anonymised datasets by the scientific community will be reviewed and determined by an independent committee within the MCRI and in accordance with institute policy.